CLINICAL TRIAL: NCT01691274
Title: A Double Blind (3rd Party Open) Randomized, Placebo Controlled, Parallel Group Dose Escalation Study To Investigate The Safety, Toleration And Pharmacokinetics Of Multiple Oral Doses Of Pf-04895162 In Healthy Subjects
Brief Title: A Study In Healthy People To Evaluate Safety, Toleration And Time Course Of Plasma Concentration Of Multiple Oral Doses Of PF-04895162
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B5311002
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Epilepsy; Phase 1; Multiple Dose; Safety; Pharmacokinetics; Toleration
MeSH Terms: conditions — Epilepsy | interventions — PF-04895162

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04895162 (Experimental)
  Interventions: Drug: PF-04895162
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04895162 — Tablets, 300 mg, single, 1 day
  Arms: PF-04895162
Drug: PF-04895162 — Tablets, 300 mg, twice a day, 14 days
  Arms: PF-04895162
Drug: PF-04895162 — Tablets, to be decided, twice a day, 14 days
  Arms: PF-04895162
Drug: Placebo — Tablets, twice a day, 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study in healthy people is to investigate safety, toleration and time course of plasma concentration of PF-04895162, following multiple oral doses for 14 days. The preliminary effect of food on Pharmacokinetics (PK) after single oral dose of PF-04895162 will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and/or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. An informed consent document signed and dated by the subject.
4. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives preceding the first dose of study medication.
* Screening supine blood pressure >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), on a single measurement (confirmed per local SOP) .
* 12 lead ECG demonstrating QTc >450 or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of <=1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Herbal supplements and hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs and postcoital contraceptive methods) and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of study medication.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* History of seizure or of a condition with risk of seizures. (A history of 1 febrile seizure in childhood does not exclude the subject.)
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | up to 12 h post dose for Days 1, 7 and 14
Time of maximum concentration (Tmax) | up to 12 h post dose for Days 1, 7 and 14
Area under the plasma concentration time profile from time zero extrapolated to inifinite time (AUCinf) | up to 12 h post dose for Days 1, 7 and 14
Area under the plasma concentration time profile from time zero to the time of last quantifiable concentration (AUClast) | up to 12 h post dose for Days 1, 7 and 14
Area under the plasma concentration time profile from time zero to quantifiable concentration 24 h post dose (AUC24) | up to 12 h post dose for Days 1, 7 and 14
AUCtau= Area under the curve from the time of dosing to the next dose (ng.hr/mL) | up to 12 h post dose for Days 1, 7 and 14
t1/2 = Terminal Elimination half life | up to 12 h post dose for Days 1, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Generaux G, Lakhani VV, Yang Y, Nadanaciva S, Qiu L, Riccardi K, Di L, Howell BA, Siler SQ, Watkins PB, Barton HA, Aleo MD, Shoda LKM. Quantitative systems toxicology (QST) reproduces species differences in PF-04895162 liver safety due to combined mitochondrial and bile acid toxicity. Pharmacol Res Perspect. 2019 Oct 9;7(6):e00523. doi: 10.1002/prp2.523. eCollection 2019 Dec. PMID 31624633
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5311002&StudyName=A%20Study%20In%20Healthy%20People%20To%20Evaluate%20Safety%2C%20Toleration%20And%20Time%20Course%20Of%20Plasma%20Concentration%20Of%20Multiple%20Oral%20Doses%20Of%20PF-048951